CLINICAL TRIAL: NCT04503525
Title: Nutritional Assessment of French Hospitalized Patients Infected With COVID-19
Brief Title: Nutritional Assessment of Hospitalized Patients With COVID-19
Acronym: DenutCOVID
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P00100
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: SARS-CoV; Nutrition Disorders
Keywords: COVID-19; Nutrition disorders
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Nutrition Disorders; COVID-19 | interventions — Nutrition Assessment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The albuminemia in blood will be determined
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID 19 hospitalized patients: COVID 19 infected patients admitted in conventional hospitalization for less than 72 hours
  Interventions: Other: Nutritional assessment

INTERVENTIONS:
Other: Nutritional assessment — Nutritional assessment in COVID patients

SUMMARY:
The nutritional consequences of the infection by the SARS-CoV-2 are as follows:

* A severe respiratory infection induces an inflammatory syndrome and hypercatabolism, as well as an increase in energy expenditure related to ventilatory work; nutritional requirements (calories and protein) are therefore increased.
* Food intake is often reduced by several factors: anorexia secondary to infection, respiratory discomfort, anosmia, ageusia, obesity, stress, confinement, organizational problems limiting meal assistance.

Then, it is important to asses the nutritional status of COVID patients hospitalized in conventional COVID units (excluding intensive care).

ELIGIBILITY:
Inclusion Criteria:

* Patient on conventional hospitalization (duration less than 72 hours)
* Age > 18 years old
* COVID 19 diagnosed by Real Time Polymerase Chain Reaction (RT-PCR)
* Patient agreed to participate in the study
* Patient affiliated to French social security

Exclusion Criteria:

* Patient hospitalized in intensive care units during more than 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with COVID 19 disease
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Nutritional status of COVID infected patients | Up to 72 hours
  The nutritional status of patients within the first 72 hours after hospital admission will be categorized according to the French Haute Authorité de Santé (France, 2019)
  * non-malnourished patient
  * moderately malnourished patient
  * severely malnourished patient

SECONDARY OUTCOMES:
Correlation between the nutritional status and the supplemental oxygen requirement | Up to 72 hours
  The supplemental oxygen requirement classified as follows:
  * non-severe: no need of Oxygen
  * light: 1 - 2 l/min
  * moderate: 3 - 5 l/min
  * severe: > 5 l/min
  * critical: mechanical ventilation
Correlation between the nutritional status and the prognostic after hospitalization | Up to 72 hours
  The prognostic after hospitalization will be classified as follows:
  * Hospital discharge
  * Transfer to the intensive care unit
  * Transfer to other unit
  * Follow-up care and rehabilitation
  * Death

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Cortet, MD, Principal Investigator — GHICL
Locations (1):
- Saint-Vincent Hospital, Lille, Haut-de-France, France

IPD SHARING:
Plan to Share IPD: No